CLINICAL TRIAL: NCT07345442
Title: A Randomized, Double-blind, Placebo-controlled, Dose Escalation Study to Assess the Safety, Tolerability, Pharmacokinetics of Single Dose and 7-day Repeat Doses of PA9159 Nasal Spray in Healthy Chinese Adult
Brief Title: Study on the Safety, Tolerability, and Pharmacokinetics of PA9159 Nasal Spray in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Palo Alto Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA9159-102
Record Dates: First submitted 2025-12-23; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Arm 1-3, the treatment is given once for one day, with escalation doses of 80 μg, 160 μg, 320 μg, After two days elution, Arm 4-6, at the escalation dose of 80 μg, 160 μg, 320 μg is given once a day for 7 days. 12 health subjects will be enrolled for each dose group, randomized proportionally at 3:1 ratio to receive either the investigational product PA9159 or placebo nasal spray, with a total of 36 subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a randomized, double-blind, placebo-controlled dose escalation phase 1 trial, including single dose and 7-day repeat doses of PA9159 nasal spray.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PA9159 80 μg single dose and placebo (Experimental): Twelve subjects will be randomly assigned at a 3: 1 ratio to receive either single dose of 80 μg PA9159 or placebo. There will be a follow-up period to review all available clinical and laboratory safety data before escalating to next dosing level.
  Interventions: Drug: PA9159 nasal spray solution, 80 μg one day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient
- PA9159 160 μg single dose and placebo (Experimental): Twelve subjects will be randomly assigned at a 3: 1 ratio to receive either single dose of 160 μg PA9159 or placebo. There will be a follow-up period to review all available clinical and laboratory safety data before escalating to next dosing level.
  Interventions: Drug: PA9159 nasal spray solution, 160 μg one day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient
- PA9159 320 μg single dose and placebo (Experimental): Twelve subjects will be randomly assigned at a 3: 1 ratio to receive either single dose of 320 μg PA9159 or placebo. There will be a follow-up period to review all available clinical and laboratory safety data.
  Interventions: Drug: PA9159 nasal spray solution, 320 μg one day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient
- PA9159 80 μg repeated doses and placebo (Experimental): Twelve subjects will be randomly assigned at a 3: 1 ratio to receive either 80 μg PA9159 or placebo once a day for 7 days. There will be follow-up period to review all available clinical and laboratory safety data before escalating to next dosing level.
  Interventions: Drug: PA9159 nasal spray solution, 80 μg 7-day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient
- PA9159 160 μg repeated doses and placebo (Experimental): Twelve Ten subjects will be randomly assigned at a 3: 1 ratio to receive either 160 μg PA9159 or placebo once a day for 7 days. There will be follow-up period to review all available clinical and laboratory safety data before escalating to next dosing level.
  Interventions: Drug: PA9159 nasal spray solution, 160 μg 7-day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient
- PA9159 320 μg repeated doses and placebo (Experimental): Twelve subjects will be randomly assigned at a 3: 1 ratio to receive either 320 μg PA9159 or placebo once a day for 7 days. There will be a follow-up period to review all available clinical and laboratory safety data.
  Interventions: Drug: PA9159 nasal spray solution, 320 μg 7-day treatment; Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient

INTERVENTIONS:
Drug: PA9159 nasal spray solution, 80 μg one day treatment — Single dose of PA9159 (20 μg/nasal spray) is delivered intranasally through a metered-dose mechanical spray pump, two sprays each in the left and right nostril.nostril.
  Arms: PA9159 80 μg single dose and placebo
Drug: PA9159 nasal spray solution, 160 μg one day treatment — Single dose of PA9159 (40 μg/nasal spray) is delivered intranasally through a metered-dose mechanical spray pump, two sprays each in the left and right nostril.
  Arms: PA9159 160 μg single dose and placebo
Drug: PA9159 nasal spray solution, 320 μg one day treatment — Single dose of PA9159 (80 μg/nasal spray) is delivered intranasally through a metered-dose mechanical spray pump, two sprays each in the left and right nostril.
  Arms: PA9159 320 μg single dose and placebo
Drug: PA9159 nasal spray solution, 80 μg 7-day treatment — Repeated doses of PA9159 (20 μg/nasal spray) or Placebo is delivered intranasally through a metered-dose mechanical spray pump, two sprays each in the left and right nostril.
  Arms: PA9159 80 μg repeated doses and placebo
Drug: PA9159 nasal spray solution, 160 μg 7-day treatment — Repeated doses of PA9159 (40 μg/nasal spray) or Placebo is delivered intranasally through a metered-dose mechanical spray pump, two sprays each in the left and right nostril.
  Arms: PA9159 160 μg repeated doses and placebo
Drug: PA9159 nasal spray solution, 320 μg 7-day treatment — Repeated doses of PA9159 (80 μg/nasal spray) is delivered intranasally through a metered-dose mechanical spray pump, two sprays each in the left and right nostril.
  Arms: PA9159 320 μg repeated doses and placebo
Drug: Placebo, the same intranasal spray solution without PA9159 active ingredient — Placebo is delivered intranasally through a metered-dose mechanical spray pump with the same volume as the corresponding PA9159 dose group

SUMMARY:
PA9159 is a highly potent novel corticosteroid. The purpose of this study is to exam the safety, tolerability, and pharmacokinetics of single and repeat dosing of intranasal PA9159, to establish maximum tolerated dose in healthy chinese adult

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled dose escalation phase 1 trial, including single dose and 7-day repeat doses of PA9159 nasal spray. In the study, the treatment is given once for one day, with escalation doses of 80 μg, 160 μg, 320 μg. After two days elution, PA9159 at the escalation dose of 80 μg, 160 μg, 320 μg is given once a day for 7 days. 12 health subjects will be enrolled for each dose group, randomized proportionally at 3:1 ratio to receive either the investigational product PA9159 or placebo nasal spray, with a total of 36 subjects for this two-part study. Subjects will be evaluated for the safety, tolerability and pharmacokinetics of PA9159 intranasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 65 years (including upper and lower limits);
* Male body weight ≥ 50 kg, female weight ≥ 45 kg, body mass index (BMI) between 19 and 26 kg/m2 (including cut-off values);
* Voluntary participation and signing of informed consent.

Exclusion Criteria:

* Those who cannot properly use a nasal spray, cannot tolerate nasal administration, or fail nasal spray administration training;
* Those with special dietary requirements who cannot adhere to a standard diet;
* Those with a history of serious diseases affecting the respiratory, cardiovascular, digestive, endocrine, hematologic, immune, or nervous systems, or currently suffering from diseases of the aforementioned systems;
* A history of recurrent (defined as more than once) or disseminated shingles, glaucoma, cataracts, or ocular infectious diseases;
* Allergic to the investigational drug or any component of the investigational drug, or having an allergic constitution (referring to being allergic to two or more foods, drugs, or environmental substances);
* Vital signs during the screening period, physical examination, nasal examination, laboratory tests (complete blood count, blood biochemistry, urinalysis, coagulation function), serum cortisol, chest X-ray, abdominal ultrasound, 12-lead electrocardiogram, and other abnormalities judged by the investigator to be clinically significant;
* Those who test positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), syphilis treponemal antibody (Syphilis TP), or HIV (HIV Ag/Ab);
* Exclude individuals who have frequently consumed alcohol in the past three months, defined as drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer with 5% alcohol, 45 mL of spirits with 40% alcohol, or 150 mL of wine with 12% alcohol), or those who tested positive on baseline breath alcohol tests, or those unable to stop alcohol intake during the study period;
* Those with a smoking history of more than 10 years, or who smoke more than 5 cigarettes per day in the 3 months prior to screening, or who cannot stop using any tobacco products during the trial, or who test positive for nicotine at baseline;
* Individuals with a history of drug abuse or drug use in the past two years, or those who tested positive for drug use in baseline urine screening;
* Individuals who have taken any medication (prescription drugs, over-the-counter drugs, Chinese herbal medicine, vaccines) or health supplements within the 2 weeks prior to screening or during the screening period;
* Exclude individuals who have used preparations containing corticosteroids or any drugs affecting CYP3A4 enzyme activity within the 30 days prior to screening or during the screening period;
* Participants who have consumed beverages or foods containing grapefruit, dragon fruit, mango, pomelo, pomegranate, papaya, or star fruit within 14 days prior to screening and during the screening period, or who do not agree to stop consuming the above foods during the trial;
* Anyone who consumes any foods or beverages rich in caffeine or methylxanthines (such as coffee, tea, cola, chocolate, seafood, cocoa, animal liver, etc.) within 48 hours prior to the first use of the investigational drug, or who does not agree to stop consuming the above foods during the trial;
* Individuals who have donated blood or experienced significant blood loss (≥400 mL) within the 90 days prior to screening, or who have used blood products or received a transfusion;
* Participants who have taken part in other clinical studies and used study products within the 90 days prior to screening;
* Individuals who have previously undergone respiratory system surgery, have had major surgery within the three months prior to screening (as determined by the investigator based on past medical history), have experienced major trauma, or plan to undergo surgery during the study period;
* Difficulty with venous blood collection, or a known history of fainting at the sight of needles or blood;
* Women who test positive for pregnancy or are breastfeeding;
* Researchers believe there are other situations in which participation in the trial is not suitable, or the subject cannot participate in the trial due to personal reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events (AEs) | up to 7 days after last nasal spray treatment
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical study subject administered a medicinal product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Pharmacokinetics of single dose and repeat doses of Nasal Spray PA9159-Cmax | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects) 0.5, 1, 1, 2, 4, 6, 8, 12,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Maximum Observed Plasma Concentration (Cmax)
Pharmacokinetics of single dose and repeat doses of Nasal Spray PA9159-Tmax | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects) 0.5, 1, 1, 2, 4, 6, 8, 12,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Time to Reach Maximum Observed Plasma Concentration (Tmax)
Pharmacokinetics of single dose and repeat doses of Nasal Spray PA9159-AUC | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects) 0.5, 1, 1, 2, 4, 6, 8, 12,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Area Under the Plasma Concentration-Time Curve (AUC)
Pharmacokinetics of single dose and repeat doses of Nasal Spray PA9159-T1/2 | Pre-dose, and post-dose (day 1 for single dose subjects, day 1 and day 7 for repeat doses subjects) 0.5, 1, 1, 2, 4, 6, 8, 12,12, 24 hours, and for repeat doses subjects, also 30 minutes pre-dose on day 4, day 5 and day 6
  Blood samples will be collected serially, and the concentrations of PA9159 in plasma samples are determined by liquid chromatography/mass spectrometry/mass spectrometry (LC/MS/MS), followed by the calculation of pharmacokinetic parameter Elimination Half-Life Period (T1/2)

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Wen, Principal Investigator — The First Affiliated Hospital of Nanchang University; Xiaohua Cheng, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No